CLINICAL TRIAL: NCT01154608
Title: Effect of Enzyme Therapy on Protein Metabolism in Chronic Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: National Research Agency, France (Other); Solvay Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Basic Science
Other Study IDs: PANCREATITE
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2010-05

CONDITIONS: Pancreatitis
Keywords: Protein absorption in pancreatitis; Protein metabolism in pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Pancrelipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pancreatic enzymes (Experimental)
  Interventions: Drug: Creon
- control (Placebo Comparator)
  Interventions: Other: No enzyme therapy

INTERVENTIONS:
Drug: Creon
  Arms: pancreatic enzymes
Other: No enzyme therapy — Current enzyme therapy of the patient is stopped during 7 days
  Arms: control

SUMMARY:
Pancreatic exocrine insufficiency is known to impair nutrient absorption, especially fat, but few data exist about protein absorption. We aimed to investigate this question and assess the enzyme substitution efficiency using a sensitive method.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pancreatitis
* Pancreatic insufficiency
* Enzyme therapy treatment

Exclusion Criteria:

* Hepatic failure
* Pregnancy
* Positive serology to HIV, HCV, AGHbS, gastro-intestinal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-04

PRIMARY OUTCOMES:
transfer of dietary nitrogen to metabolic pools

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche sur Volontaires, Bobigny, France